CLINICAL TRIAL: NCT02691988
Title: Withdrawal of Inhaled Corticosteroids and the Possible Effect on Exacerbation Rate in Primary Care Patients With COPD
Brief Title: Withdrawal of Inhaled Corticosteroids in Primary Care Patients With COPD
Acronym: WHISPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Novartis (Industry); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL52880.091.15
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Inhaled corticosteroids; General practice; Primary care; Pharmacotherapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICS withdrawal (Experimental): Guided ICS withdrawal combined with optimization of bronchodilator treatment
  Interventions: Other: ICS withdrawal
- Usual care (Active Comparator): Optimization of bronchodilator treatment
  Interventions: Other: Usual care

INTERVENTIONS:
Other: ICS withdrawal — Bronchodilator therapy is optimized according to the latest COPD guideline of the Dutch College of General Practitioners (NHG) and inhaled corticosteroids are withdrawn.
  Arms: ICS withdrawal
Other: Usual care — Bronchodilator therapy is optimized according to the latest COPD guideline of the Dutch College of General Practitioners (NHG)
  Arms: Usual care

SUMMARY:
Rationale: Because long-term use of ICS is associated with an increased likelihood of side-effects such as increased risk of pneumonia and loss of bone density, it is important to limit prescription of ICS to patients who have a clear indication for this treatment. In addition, avoiding unnecessary treatment with ICS could reduce the burden that chronic obstructive pulmonary disease (COPD) puts on healthcare budgets. The recently updated COPD guideline of the Dutch college of General Practitioners (NHG) emphasizes the importance of optimizing medical treatment for COPD patients with only limited room for the use of inhaled corticosteroids.

Objective: The objective of the study is to investigate whether discontinuation of inhaled corticosteroids (ICS) for patients without a clear indication for ICS according to current guidelines results in a reduction of ICS use without adverse health effects for the patients involved.

Study design: The study is a pragmatic, clustered, parallel group, non-inferiority trial in Dutch general practices with a follow-up of 26 weeks per patient.

Study population: 620 COPD patients with confirmed chronic airflow obstruction, aged ≥ 40 yrs who use ICS for at least the prior 6 months without a clear indication.

Intervention (if applicable): Guided ICS withdrawal in optimised COPD management. All study participants (of both study arms) will receive recommendations on optimal bronchodilator therapy and a personalized action plan to recognize symptom deterioration in an early stage.

Main study parameters/endpoints: Number of exacerbation-free weeks. Secondary study parameters: successful cessation of ICS, time to first exacerbation, number of moderate and severe exacerbations, health-related quality of life, health status, and pneumonias. Moreover, information on the process of care and costs will be collected.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Many COPD patients use ICS without a clear indication. Long-term use of ICS is associated with an increased likelihood of side-effects such as increased risk of pneumonia and loss of bone density and should be avoided in those who do not benefit from it. However, there is a small subgroup of COPD patients that have reduced numbers of exacerbations because of their ICS use and it is impossible to identify a priori the patients who this applies too. Therefore, it is important that the ICS discontinuation is guided to detect potential deteriorations early on.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis in the medical record (ICPC code R95 or R91);
* Most recent spirometry result is less than three years old and shows a ratio of the Forced Expiratory Volume in 1 second (FEV1) to the Forced Vital Capacity (FVC) of less than 0.7, in short: FEV1/FVC ratio <0.7 (If no recent spirometry results are available, the patient will be scheduled for a diagnostic spirometric test);
* ICS treatment for at least the past 6 months;
* Accessible electronic medical record and prescription data history of at least one year;
* The subject's COPD is primarily managed by the general practioner (GP) (i.e., not by a chest physician); or if a subject's COPD is treated by a chest physician as well, the chest physician agrees with the invitation of the subject.
* Willing to provide written informed consent;
* Mentally competent.

Exclusion Criteria:

* A spirometry test that has demonstrated airflow reversibility (i.e., post-bd FEV1 improvement of at least 12% and 200 ml compared to baseline and/or post-bd FEV1 improvement of 9% of the baseline FEV1 % predicted value) that preceded the initiation of ICS treatment;
* Diagnosis of asthma in the medical record (ICPC code R96);
* Allergic respiratory disease which has been confirmed by a positive skin prick test or specific immunoglobulin E (IgE) in serum as documented in the medical record, in combination with a documented history respiratory allergic symptoms;
* Two or more exacerbations in the previous 12 months that were treated with oral corticosteroids, antibiotics, or both; and/or required a visit to an emergency care facility or hospital admission;
* Use of oral corticosteroids on a regular basis (i.e., more than six weeks in the previous half year) for any reason;
* Currently participating in another intervention study that interferes with the current study;
* Has one or more serious other diseases that are likely to lead to study drop-out (e.g., diseases with limited life expectancy) or influence the study results; or
* Pregnancy or women who are trying to conceive a child;
* Unable to read or understand the Dutch language.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of exacerbation-free weeks (EFWs) | 6 months
  Weeks in which the patient does not experience a worsening of his respiratory condition according to accepted symptom-based definitions of an exacerbation. This outcome is measured on a weekly basis with the Telephonic Exacerbation Assessment System (TEXAS)

SECONDARY OUTCOMES:
Successful ICS withdrawal | 6 months
  The proportion of patients with successful cessation of ICS, i.e. a period of 26 weeks after the withdrawal date without the occurrence of a moderate or severe exacerbation or reintroduction of ICS treatment.
Time to first exacerbation | Max. 6 months
  Time (in weeks) to first exacerbation will be calculated for all subjects. The definition for an exacerbation will be comparable to the definition used for EFWs. Information on time to first exacerbation will be collected using TEXAS.
Moderate and severe exacerbations | 6 months
  A moderate exacerbation is defined as prescription of a course of oral corticosteroids and/or antibiotics related to deterioration of COPD registered as episodes in the electronic patient record. A severe exacerbation is defined as a COPD-related ER visit and/or unscheduled COPD-related hospital admission.
Health status (CCQ) | 6 months
  Health status will be measured using the Clinical COPD Questionnaire (CCQ) which has been developed as a COPD specific health status measurement. CCQ questionnaires that are filled out at the start (t=0) and end of the study period (t = 26 weeks) will be used to evaluate the difference in change in CCQ score between the intervention and control groups.
Health-related quality of life (HRQoL) | 6 months
  Disease specific HRQoL will be assessed with the Short-form Chronic Respiratory Questionnaire (SF-CRQ) at baseline and 26 weeks of follow up.
General health state (EQ-5D-3L) | 6 months
  The EuroQol-5 Dimensions-3 Levels (EQ-5D-3L) will be used to assess the general health state of subjects at the start and after 26 weeks.
Side effects of inhaled corticosteroids | 6 months
  Side effects of inhaled corticosteroids will be measured using the Inhaled Corticosteroids Questionnaire Short form (ICQ-S).

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Centre, Department of Primary and Community Care, Nijmegen, Netherlands